CLINICAL TRIAL: NCT06455020
Title: Catheter Ablation of Haemodynamically Not-tolerated Electrical Storm in Structural Heart Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-vtstorm
Record Dates: First submitted 2024-06-07; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Ventricular Tachycardia
Keywords: Catheter ablation; Mortality; Electrical storm
MeSH Terms: conditions — Tachycardia, Ventricular | interventions — Catheter Ablation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Catheter ablation (Experimental): Patients randomized to the emergency catheter ablation arm will first undergo catheter ablation. Vasopressors, antiarrhythmic drugs, and hemodynamic mechanical support devices will be adopted as needed. All patients will be advised for ICD implantation before discharge.
  Interventions: Procedure: Catheter ablation
- Stepped-care strategies (Active Comparator): Patients randomized to the stepped-care strategies arm will undergo a stepwise progressive procedure, with anti-arrhythmic drugs, sedation and anesthesia, and hemodynamic mechanical support devices, that is, the next treatment is only started when the previous sequence of treatment is ineffective, and catheter ablation is only used as the final rescue treatment. All patients will be advised for ICD implantation before discharge.
  Interventions: Procedure: Stepped-care strategies

INTERVENTIONS:
Procedure: Catheter ablation — Emergency catheter ablation is defined as ablation performed within 48 hours of hospital admission
  Arms: Catheter ablation
Procedure: Stepped-care strategies — Patients randomized to the stepped-care strategy arm will receive treatment through a systematic, stepwise protocol beginning with anti-arrhythmic drugs, followed by sedation and anesthesia, and progressing to haemodynamic mechanical support devices if earlier treatments prove ineffective. Catheter ablation will be reserved as the final rescue intervention.
  Arms: Stepped-care strategies

SUMMARY:
This is a multi-center, parallel-group, randomized, open-label trial evaluating the clinical outcome and efficacy of emergency catheter ablation versus conventional stepped-care strategies in patients with haemodynamically not-tolerated ventricular tachycardia (VT).

DETAILED DESCRIPTION:
The prognosis of haemodynamically not-tolerated VT in structural heart disease is very poor, with a high 30-day mortality rate >30%, resulting in extremely heavy medical burden. Current guidelines lack specific recommendations for managing this condition. The prevailing treatment strategy involves a sequential approach-beginning with anti-arrhythmic drugs, sedation, and anesthesia, followed by haemodynamic mechanical support devices. Catheter ablation is only used as the final rescue treatment. Typically, patients undergo repeated electrical cardioversion and receive multiple vasopressors and antiarrhythmic drugs, facing increased risks of complications from enhanced haemodynamic support. Studies have shown that these patients often eventually progress to irreversible pump failure, miss the window for effective catheter ablation, and ultimately die. Early cardioversion and maintenance of sinus rhythm, may significantly reduce mortality rates in patients with haemodynamically not-tolerated VT. Therefore, emergency catheter ablation is expected to reduce the mortality of haemodynamically not-tolerated ventricular tachycardia.

In this study, we aim to evaluate the effect of emergency catheter ablation in haemodynamically not-tolerated ventricular tachycardia. Current study will include 96 patients, and all patients will be randomized to either the emergency catheter ablation arm or stepped-care strategies arm in a 1:1 fashion. The follow-up duration is 1 year. The primary outcome is a composite outcome of VT recurrence, cardiovascular re-hospitalization, and all-cause mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 80 years;
2. Having structural heart disease, including ischemic cardiomyopathy and nonischemic cardiomyopathy;
3. Haemodynamically not-tolerated, defined as persistent hypotension (systolic blood pressure <90 mmHg and mean arterial pressure 30 mmHg lower than baseline or <70 mmHg, with associated signs of end-organ hypoperfusion);
4. Electrical storm, defined as >3 VT episodes within 24 hours.

Exclusion Criteria:

1. Reversible causes of ventricular tachycardia or cardiomyopathy;
2. Ventricular thrombosis diagnosed by echocardiography and/or cardiac magnetic resonance;
3. Acute ST-segment-elevation myocardial infarction within 60 days;
4. Cardiac surgery within 60 days;
5. Unstable angina;
6. Pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Composite outcomes of ventricular tachycardia recurrence, cardiovascular hospitalization, or death during the 30-day follow-up | 30 days
  Recurrent ventricular tachycardia is defined as any appropriate implantable cardiac defibrillation therapy (shock or antitachycardia pacing) or documented sustained monomorphic ventricular tachycardia >30 seconds. Cardiovascular rehospitalization is defined as a hospital admission after the randomly assigned procedure for heart failure, procedure-associated complications, or arrhythmic causes during the 30-day follow-up.

SECONDARY OUTCOMES:
Recurrence of ventricular tachycardia during the 30-day follow-up | 30 days
  Recurrent ventricular tachycardia is defined as any appropriate implantable cardiac defibrillation therapy (shock or antitachycardia pacing) or documented sustained monomorphic ventricular tachycardia >30 seconds during the 30-day follow-up.
Cardiovascular re-hospitalization during the 30-day follow-up | 30 days
  Cardiovascular re-hospitalization is defined as a hospital admission after the randomly assigned procedure for heart failure, procedure-associated complications, or arrhythmic causes during the 30-day follow-up.
All-cause mortality during the 30-day follow-up | 30 days
  All-cause mortality is defined as the death from all causes during the 30-day follow-up.
Composite outcomes of ventricular tachycardia recurrence, cardiovascular hospitalization, or death during the 1-year follow-up | 1 year
  Recurrent ventricular tachycardia is defined as any appropriate implantable cardiac defibrillation therapy (shock or antitachycardia pacing) or documented sustained monomorphic ventricular tachycardia >30 seconds. Cardiovascular rehospitalization is defined as a hospital admission after the randomly assigned procedure for heart failure, procedure-associated complications, or arrhythmic causes during the 1-year follow-up.
All-cause mortality during the 1-year follow-up | 1 year
  All-cause mortality is defined as the death from all causes during the 1-year follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Deyong Long, MD, Principal Investigator — Beijing Anzhen Hospital
Locations (4):
- China (4):
  - Beijing Anzhen Hospital, Capital Medical University, Beijing
  - Second Xiangya Hospital, Central South University, Changsha
  - The Affiliated YanAn Hospital of KunMing Medical University, Kunming
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing

IPD SHARING:
Plan to Share IPD: No